CLINICAL TRIAL: NCT04416126
Title: A Phase 1 Randomized, Double Blinded, Placebo Controlled, Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single Doses of ARCT-810 in Healthy Adult Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of ARCT-810 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARCT- 810-01
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Ornithine Transcarbamylase Deficiency
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded, Placebo Controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARCT-810 (Experimental): Ascending single doses of ARCT-810 administered intravenously
  Interventions: Biological: ARCT-810
- Placebo (Placebo Comparator): Single doses of 0.9% Saline administered intravenously
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARCT-810 — ARCT-810 is an investigational medicinal product comprising OTC mRNA formulated in a lipid nanoparticle (LNP) under development.
  Arms: ARCT-810
Other: Placebo — The placebo for this study is 0.9% sterile saline.
  Arms: Placebo

SUMMARY:
Determine the safety, tolerability and pharmacokinetics of single doses of ARCT-810 in healthy adult subjects.

DETAILED DESCRIPTION:
This is a single ascending dose study of ARCT-810 in which approximately 30 subjects are planned to be enrolled. The length of each study participant is approximately 8 weeks from screening to last study visit.

Study participants will be allocated to one of the five different study groups (also called cohorts), to test different doses of ARCT-810. There will be 6 participants in each group. Within each cohort, subjects will be randomized 2:1 to receive ARCT-810 or placebo as an IV infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged 18 to 65 at the time of informed consent.
2. Body weight ≤ 100Kg and body mass index <35 kg/m2
3. Willing to refrain from strenuous exercise/activity (for example heavy lifting, weight training, intense aerobics classes etc.) and alcohol for at least 72 hours prior to study visits and willing to refrain from taking protein supplements for the duration of the study.
4. Willing and able to comply with protocol-defined procedures and complete all study visits
5. Males must be surgically sterile or, if engaged in sexual relations with a female of child-bearing potential, the subject must be using an acceptable contraceptive method from the time of signing the informed consent form until at least 30 days after the last dose of Study Drug. Females: must be non-pregnant and non-lactating and either: i. surgically sterile or ii. post-menopausal

Exclusion Criteria:

1. Clinically significant abnormalities in medical history
2. Screening laboratory results as follows:

   * ALT, AST, GGT, total bilirubin or alkaline phosphatase, > ULN.
   * Random blood glucose and/or HbA1c > ULN
   * Hemoglobin < LLN
   * Platelet count < 100x109/L
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 calculated by Modification to Diet in Renal Disease [MDRD] study equation.
   * Urine protein:creatinine ratio (UPCR) > 50 mg/mmol
3. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed within 7 days prior to Study Day 1
4. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
5. Uncontrolled hypertension (BP > 160/100 mm Hg)
6. Treatment with another investigational drug, biological agent, or device within one month of screening, or 5 half-lives of investigational drug, whichever is longer
7. Recent (within 1 year) history of, or current drug or alcohol abuse
8. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the Study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and dose-relationship of AEs | 4 weeks
  Safety and tolerability of ARCT-810 assessed by determining the incidence, severity and dose-relationship of AEs by dose

SECONDARY OUTCOMES:
Number of participants with changes in plasma pharmacokinetic parameters after single dose of ARCT-810 | Up to 15 days
  The plasma pharmacokinetics (concentration-time results) of ARCT-810 will be assessed following single dose
Number of participants with changes in urine pharmacokinetic parameters after single dose of ARCT-810 | Up to 24 hours
  The urine pharmacokinetics (concentration-time results) of ARCT-810 will be assessed following single dose

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schwabe, MD, Principal Investigator — Auckland Clinical Studies (ACS) Ltd.
Locations (1):
- Auckland Clinical Studies (ACS) Ltd., Auckland, New Zealand